CLINICAL TRIAL: NCT06217575
Title: BRAIN-SPEED-VETS: Brain Research Assessing Impacts of Neurophysiological Processing Speed Training in Veterans
Brief Title: Brain Research Assessing Impacts of Neurophysiological Processing Speed Training in Veterans
Acronym: BRAIN-SPEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Birmingham VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Keith McGregor, Associate Professor, Birmingham VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300011767
Record Dates: First submitted 2023-12-14; First posted 2024-01-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury; Aging; Cognitive Decline
Keywords: cognitive decline; visual attention training; useful field of view; mild traumatic brain injury; aging
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Cognitive Dysfunction | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Attention Training (Active Comparator): Visual attention training is at the core of well-known training programs such as useful field of view (UFOV) training. The adapted nature of the computerized training approach affords individual differences in performance at the training outset while evaluating gains using specified performance criteria. Training parameters (duration of stimulus presentation for processing speed) are adjusted based on accuracy.
  Interventions: Behavioral: Visual Attention Training
- Alpha Neurofeedback training (Experimental): Electroencephalogram (EEG) based neurofeedback (NFB) is a method in which brain activity is modulated via self-induced increases or decreases in the power of selected EEG frequency bands. The subject's control over his or her EEG activity is mediated with visual feedback. We will employ alpha neurofeedback training to examine how this conditioning paradigm may improve visual attention.
  Interventions: Behavioral: Alpha neurofeedback training

INTERVENTIONS:
Behavioral: Alpha neurofeedback training — Alpha neurofeedback training affords the participant the ability to monitor cortical EEG waves and entrain to a specific rhythm using visual feedback. Alpha is measured between 8-12Hz and is associated with cortical inhibition. Aging related changes in alpha have been associated with loss of modulation ability. However, alpha training may afford increased perception of visual details.
  Other Names: alpha modulation; neurofeedback; eeg-nfb
  Arms: Alpha Neurofeedback training
Behavioral: Visual Attention Training — Visual attention training involves repeated testing on the location and identity of objects in the visual field. Also called the "Dual Decision" task training, objects are briefly presented in a radial field of view surrounding a gaze fixation point. The participant is asked to remember the location and object presented within the field. The test progressively increases in difficulty by limiting the amount of time the object is presented on screen. Accuracy is measured by either a correct or incorrect response (binary response).
  Other Names: Standard Visual Attention Training; dual decision
  Arms: Visual Attention Training

SUMMARY:
Older veterans with a history of mild brain trauma exhibit early cognitive challenges, especially in driving-related tasks. This is attributed to alterations in the brain's excitatory/inhibitory (E/I) balance. This pilot project investigates this phenomenon by leveraging electroencephalography (EEG) to measure parietal lobe alpha rhythms during visual attention tasks. The hypothesis is that targeted visual attention training can modulate these alpha rhythms, improving instrumental activities in daily life. However, outcomes from such training vary, possibly due to individual differences in cortical inhibitory functions. This study will assess the relationship between EEG measures of E/I balance pre- and post-visual attention training and its effects on processing speeds in aging veterans. Our findings aim to provide a foundation for customized therapies and interventions for veterans with and without a history of brain trauma.

DETAILED DESCRIPTION:
Veterans aged 50 and above who have suffered mild traumatic brain injury (mTBI) are twice as prone to develop dementia. From 2001, during the Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) campaigns, over 470,000 veterans were diagnosed with TBI. Beyond the prevalence of the signature wound of the OEF and OIF campaigns, the number of mTBI cases within the VA system is believed to be much higher. Disturbingly, an increasing number of veterans, especially those with TBI, are being diagnosed with mild cognitive impairment and frank dementia between ages 50-60. With 72% of veterans (13.2 million, a figure rising yearly) over 50 years old (Vetpop, 2020), the VA needs to implement preventative and rehabilitative interventions to limit the growing impact of cognitive decline in the veteran population.

Cognitive training paradigms have been developed and tested over the past decades, with some controversy over the overall effect10. Programs such as repeated task practice (e.g., list memorization and mnemonics) have shown mixed results in aggregate, primarily due to a lack of training transfer across domains. In contrast, process-based cognitive training has consistently improved general cognitive ability with one program, visual attention training, showing considerable transfer effects. Also known as speed-of-processing training (cf. - useful field-of-view [UFOV]), visual attention training is done on a computer and targets perceptual deficits associated with aging and TBI.

Changes in brain function that reduce the ability for perceptual information to be processed are likely mechanisms of impaired cognition. Visual attention training was developed to increase visual perception directly to counteract deficient visual fields. Previous studies have shown that visual attention training increases instrumental daily activities pertinent to driving performance, resulting in prolonged driving mobility. Unfortunately, visual attention training paradigms have required an extended training duration (months) and tend to show varied outcomes. The identified cognitive mechanism of increased perceptual detail processing is quite powerful, but individual training response may depend on one's ability to apply selective cortical inhibition. Cortical oscillations measured with electroencephalography (EEG) are believed to reflect such inhibition. Recent EEG work during visual attention training has shown that people exhibiting selective engagement of alpha patterns have faster processing speed and better perceptual discrimination.

Our recent VA-funded projects in aging have shown that procedural motor learning performance is related to individual differences in excitatory/inhibitory (E/I balance) assessed with transcranial magnetic stimulation (TMS) (Novak et al., under review). Moreover, recent work has also shown that neurological changes in cortical activity are evident after just 10 hours of visual attention training. The current project will evaluate changes in EEG measures of cortical inhibition in older veterans to improve perceptual processing using an adapted visual attention training program. The present work expands on prior work in neuromodulation using low-cost, nonpharmacological rehabilitation techniques.

ELIGIBILITY:
Inclusion Criteria:

Ages: 18-35 (Younger Group); Ages 50-80 (Healthy Older Group); Ages 50-85 (persons with a history of mild traumatic brain injury)

* English speaking
* Veterans with mild traumatic brain injury (mTBI):
* A history of mTBI confirmed by the Ohio State University TBI Identification Method-Short Form (including a requirement that the mTBI caused a loss of consciousness lasting less than 30 min).
* An additional note will be made for Veterans with mTBI with a report of objective or subjective cognitive decline not meeting the criteria (i.e.- Montreal Cognitive Assessment (MoCA) >23) for impairment

Exclusion Criteria:

Failure to provide informed consent

* Metal of foreign objects in the body that would interfere with an magnetic resonance imaging (MRI) or transcranial magnetic stimulations (TMS)
* History of penetrating head wounds or a diagnosis of moderate/severe TBI
* Participants with significant visual field deficits were excluded, as were those with active suicidal ideation

  * Suicidal ideation will be assessed with the Columbia suicidality scale (C-SSRS)
  * Participants with active ideation will be referred to the Veteran Crisis Line (988) (or walked) to the Front Door program at the Birmingham East clinic
* Participation in a concurrent clinical trial that could affect study outcome (however, participation in standard treatments e.g. occupational therapy or use of prescribed medications such as antidepressants is acceptable)
* Smoker > 1 pack per day
* Significant cognitive impairment defined as <23 on Montreal Cognitive Assessment (MoCA) or diagnosis of mild cognitive impairment or dementia
* Visual (corrected acuity <20/80) and motor capacity (completion of 9-hole pegboard) to use a computerized intervention
* In-patient status
* Severe visual impairment, which would preclude completion of the assessments
* Progressive, degenerative neurologic disease, e.g., Parkinsons Disease, multiple sclerosis
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement Actively taking GABAergic agonist/antagonist medication (benzodiazepines, gabapentin, etc.)
* Terminal illness with a life expectancy of less than 12 months, as determined by a physician
* Other significant co-morbid diseases that would impair the ability to participate, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar disorder, schizophrenia), heavy alcohol use (>15 drinks per week); persons with depression will not be excluded
* Unable to communicate because of severe hearing loss, speech disorder or language barrier

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Specific domains of cognitive function | 6 weeks
  Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter.

SECONDARY OUTCOMES:
General Cognitive function | 6 weeks
  General cognitive function assessed by the Montreal Cognitive Assessment (MoCA) test on a scale of 0-30 points. Scores are interpreted as follows: >26 indicates no dementia, 18-26 mild cognitive impairment, 6-10 moderate dementia, and <6 severe dementia.
Quality of life as measured by SF-12 | 6 Weeks
  Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).

CONTACTS AND LOCATIONS:
Locations (1):
- CH19 933 19th St S, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No